

Document Date: June 23, 2022

# Three Dimensional Assessment of Maxillary Molars Following Distalization Using Two Different Approaches

A Thesis
Submitted to Faculty of Dentistry
Ain-Shams University
In Partial Fulfillment of the Requirements of
Master's Degree in Orthodontics

Faculty of Dentistry Ain Shams University 2022

# Statistical analysis

Statistical analysis was performed with SPSS  $20^{\mathbb{R}_*}$ , Graph Pad Prism $^{\mathbb{R}^{**}}$ , and Microsoft Excel  $2016^{***}$ .

All quantitative data were explored for normality by using Shapiro Wilk Normality test and presented as means and standard deviation (SD) values. All qualitative data were presented as frequency & percentage. All data were presented in (43) tables & (38) graphs.

#### Tests used:

- Comparisons 2 different groups was performed by using <u>Mann Whitney</u> test.
- Comparisons 2 successive follow ups periods was performed by using Paired t-test.
- Comparison between quantitative continuous data (Age & Duration) was performed by <u>Independent t-test</u>.
- Comparison between qualitative dichotomous data (Gender) was performed by <u>Chi square test</u>.
- Reliability test was performed by using <u>Intra-class Correlation Coefficient</u>
  (ICC).

<sup>\*</sup> Statistical Package for Social Science, IBM, Armonk, NY, USA.

<sup>\*\*</sup> Graph Pad Technologies, San Diego, CA, USA

<sup>\*\*\*</sup> Microsoft Co-operation, Redmond, WA, USA.

#### \* All results presented as:

- I. Normality test.
- II. Baseline characteristics:
  - A. Age.
  - B. Gender.
  - C. Duration
  - D. Pretreatment measurements. (Appendix IV).

#### III. Measurements

# The following measurements were carried for both group I and group II as well as in comparison between the two groups.

- A. Skeletal measurements
  - 1. Skeletal antero-posterior measurements.
  - 2. Skeletal vertical measurements.
- B. Dental measurements
  - 1. Angular
  - 2. Linear
- C. Soft tissue measurements.
- IV. Reliability: (Appendix V)
  - A. Inter-observer.
  - B. Intra-observer.

#### I. Normality test:

Exploration of the given data was performed using Shapiro-Wilk test and Kolmogorov-Smirnov test for normality. As Listed in (**Table 11**) and showed in (**Figure 53**), it was revealed that the significant level (P-value) was shown to be insignificant as P-value > 0.05, which indicated that alternative hypothesis was rejected, and the concluded data originated from normal distribution (parametric data) resembling normal Bell curve in pre & post measurements while P value was significant in the difference between both groups which indicated nonparametric data.

Table (11): Normality exploration of both groups regarding all measurements:

| Measur | rements | Group I<br>Single Coil Spring | Group II<br>Double Coil Spring |
|---|---|---|---|
| | Pre | > 0.05 | > 0.05 |
| Skeletal. | Post | > 0.05 | > 0.05 |
| | Difference | < 0.05* | < 0.05* |
| | Pre | > 0.05 | > 0.05 |
| Dental | Post | > 0.05 | > 0.05 |
| | Difference | < 0.05* | < 0.05* |
| | Pre | > 0.05 | > 0.05 |
| Soft tissue | Post | > 0.05 | > 0.05 |
| | Difference | < 0.05* | < 0.05* |

<sup>\*</sup> Significant difference as P < 0.05





Figure (53): Scattered chart represents normal bell curve of normality test.

#### II. Baseline characterized:

#### 1. **Age:**

In group I, minimum age was (18.4), maximum was (21.2), while mean  $\pm$  standard deviation was (19.42  $\pm$  1.03). In group II, minimum age was (18.08), maximum was (23.17), while mean  $\pm$  standard deviation was (20.7  $\pm$  2.24), as presented in table (12) and figure (54).

Comparison between both groups was performed by using Independent t-test which revealed insignificant difference between them as P > 0.05, as presented in table (12).

Table (12): Minimum, maximum, mean & standard deviation of age in both groups:

| | Min | Max | M | SD | P value |
|------|-------|-------|-------|------|---------|
| GI | 18.4 | 21.2 | 19.42 | 1.03 | 0.09 |
| G II | 18.08 | 23.17 | 20.7 | 2.24 | 0.09 |

N: count Min: minimum Max: maximum

M: mean SD: standard deviation



Figure (54): Bar chart showing mean of age in both groups.

#### 2. Gender:

In gender all companions were performed by using Chi square test. In group I, male (16.67%) was significantly lower than female (83.3%) as P < 0.05, while in group II male (33.3%) was insignificantly lower than female (66.6%) as P > 0.05, as presented in table (13) and figure (55).

Also, comparison between group I & II reveled insignificant difference between them in both male & female as P > 0.05 as presented in table (13).

<u>Table (13): Frequency & percentage of gender distribution in both</u> groups:

| Group | Ma | ale | Fen | P value | |
|----------|----|--------|-----|---------|---------|
| Group | N | % | N | % | 1 value |
| Group I | 2 | 16.67% | 10 | 83.33% | 0.001* |
| Group II | 3 | 33.33% | 6 | 66.67% | 0.13 |
| P value | 0 | 34 | 0. | | |

N: count %: percentage



**Figure (55):** Bar chart showing percentage of gender distribution in both groups

#### 3. **Duration:**

In group I, minimum duration was (5.5 months), maximum was (9.73 months), while mean  $\pm$  standard deviation was (8.03  $\pm$  2.9). In group II, minimum duration was (4 moths), maximum was (14.9 months), while mean  $\pm$  standard deviation was (10.59  $\pm$  3.89).

Comparison between both groups was performed by using Independent t-test which revealed insignificant difference between them as P>0.05, as presented in table (14) and figure (56).

<u>Table (14): Minimum, maximum, mean & standard deviation of</u> duration in months in both groups:

| | Min | Max | M | SD | P value |
|----------|------|-------|-------|------|---------|
| Group I | 5.50 | 9.73 | 8.03 | 2.90 | 0.00 |
| Group II | 4.00 | 14.90 | 10.59 | 3.89 | 0.09 |

M: mean SD: standard deviation



Figure (56): Bar chart showing mean of duration in months in both groups.

# **III.** Measurements:

# A. Skeletal:

#### 1. Anteroposterior:

#### • Group I:

In group I pretreatment records, post treatment records and difference between them regarding anteroposterior skeletal measurements were presented in table (15) and figure (57).

Comparison between pretreatment & post treatment records was performed by using Paired t-test which revealed insignificant difference between them in all measurements as P > 0.05, as presented in table (15).

Table (15): Mean & standard deviation of pretreatment, post treatment records and difference between them regarding anteroposterior skeletal measurements in group I:

| Group I<br>Anteroposterior | Pre | | Post | | Difference | | P value |
|---|---|---|---|---|---|---|---|
| Skeletal<br>Measurements | M | SD | M | SD | M | SD | 1 value |
| SNA angle | 83.41 | 4.33 | 83.47 | 3.90 | 0.05 | 1.26 | 0.854 |
| SNB angle | 77.98 | 3.18 | 77.44 | 2.53 | -0.54 | 1.36 | 0.194 |
| ANB angle | 5.50 | 2.11 | 6.07 | 2.53 | 0.57 | 1.72 | 0.273 |
| A-NV distance | 6.79 | 4.69 | 6.96 | 3.87 | 0.17 | 1.11 | 0.611 |
| Pog-NV distance | 6.06 | 6.44 | 6.02 | 5.32 | -0.04 | 2.20 | 0.951 |

M: mean SD: standard deviation



**Figure (57):** Bar chart showing mean of pretreatment, post treatment records and difference between them regarding anteroposterior skeletal measurements in group I.

# • Group II:

In group II pretreatment records, post treatment records and difference between them regarding anteroposterior skeletal measurements were presented in table (16) and figure (58).

Comparison between pretreatment & post treatment records was performed by using Paired t-test which revealed insignificant difference between them in all measurements as P > 0.05, as presented in table (16).

Table (16): Mean & standard deviation of pretreatment, post treatment records and difference between them regarding anteroposterior skeletal measurements in group II:

| Group II<br>Anteroposterior | Pre | | Post | | Difference | | r P value |
|---|---|---|---|---|---|---|---|
| Skeletal<br>Measurements | M | SD | M | SD | M | SD | P value |
| SNA angle | 83.64 | 4.14 | 83.62 | 4.15 | -0.02 | 1.07 | 0.952 |
| SNB angle | 79.27 | 3.08 | 79.13 | 3.03 | -0.14 | 1.24 | 0.735 |
| ANB angle | 4.36 | 1.72 | 4.49 | 1.63 | 0.12 | 0.54 | 0.517 |
| A-NV distance | 7.44 | 3.13 | 7.09 | 3.00 | -0.35 | 0.74 | 0.195 |
| Pog-NV distance | 8.10 | 3.71 | 7.31 | 3.26 | -0.79 | 2.04 | 0.277 |

M: mean SD: standard deviation



**Figure (58):** Bar chart showing pretreatment, post treatment records and difference between them regarding anteroposterior skeletal measurements in group II.

#### • Comparison between both groups:

Comparison between group I & II regarding difference between pretreatment & posttreatment records of anteroposterior skeletal measurements was performed by using Mann Whitney test which revealed insignificant difference between them regarding all measurements, as presented in table (17) and figure (59).

Table (17): Comparison between both groups regarding anteroposterior skeletal measurements:

| Difference | Gro | up I | Gro | Dureline | |
|---|---|---|---|---|---|
| Anteroposterior Skeletal Measurements | MD | SD | MD | SD | P value |
| SNA angle | 0.05 | 1.26 | -0.02 | 1.07 | 0.81 |
| SNB angle | -0.54 | 1.36 | -0.14 | 1.24 | 0.75 |
| ANB angle | 0.57 | 1.72 | 0.12 | 0.54 | 0.75 |
| A-NV distance | 0.17 | 1.11 | -0.35 | 0.74 | 0.24 |
| Pog-NV distance | -0.04 | 2.20 | -0.79 | 2.04 | 0.11 |

MD: mean difference

SD: standard deviation



**Figure (59):** Bar chart showing comparison between both groups regarding anteroposterior skeletal measurements.

#### 2. Vertical:

#### • Group I:

In group I pretreatment records, post treatment records and difference between them regarding vertical skeletal measurements were presented in table (18) and figure (60).

Comparison between pretreatment & post treatment records was performed by using Paired t-test which revealed insignificant difference between them in all measurements as P > 0.05, as presented in table (18).

Table (18): Mean & standard deviation of pretreatment, post treatment records and difference between them regarding vertical skeletal measurements in group I:

| Group I<br>Vertical | Pi | Pre | | Post | | rence | |
|---|---|---|---|---|---|---|---|
| Skeletal<br>Measurements | M | SD | M | SD | MD | SD | P value |
| PP-SN angle | 8.66 | 3.09 | 8.96 | 3.81 | 0.31 | 0.91 | 0.425 |
| ANS-Me distance | 63.77 | 4.78 | 63.81 | 5.66 | 0.04 | 1.43 | 0.924 |
| MP-SN angle | 36.91 | 4.09 | 36.76 | 4.20 | -0.15 | 0.61 | 0.265 |

M: mean SD: standard deviation MD: mean difference



**Figure (60):** Bar chart showing mean of pretreatment, post treatment records and difference between them regarding vertical skeletal measurements in group I.

#### • Group II:

In group II pretreatment records, post treatment records and difference between them regarding vertical skeletal measurements were presented in table (19) and figure (61).

Comparison between pretreatment & post treatment records was performed by using Paired t-test which revealed insignificant difference between them in all measurements as P > 0.05, as presented in table (19).

Table (19): Mean & standard deviation of pretreatment, post treatment records and difference between them regarding vertical skeletal measurements in group II:

| Group II<br>Vertical | Pre | | Post | | Difference | | P value |
|---|---|---|---|---|---|---|---|
| Skeletal<br>Measurements | M | SD | M | SD | MD | SD | r value |
| PP-SN angle | 9.47 | 3.58 | 9.64 | 3.31 | 0.17 | 0.27 | 0.54 |
| ANS-Me distance | 65.55 | 4.86 | 65.04 | 5.93 | -0.52 | 1.66 | 0.376 |
| MP-SN angle | 36.99 | 3.05 | 36.55 | 2.81 | -0.44 | 1.40 | 0.377 |

M: mean

SD: standard deviation

MD: mean difference



**Figure (61):** Bar chart showing mean of pretreatment, post treatment records and difference between them regarding vertical skeletal measurements in group II.

#### Comparison between both groups:

Comparison between group I & II regarding difference between pretreatment & posttreatment records of vertical skeletal measurements was performed by using Mann Whitney test which revealed insignificant difference between them regarding all measurements, as presented in table (20) and figure (62).

<u>Table (20): Comparison between both groups regarding vertical skeletal</u> measurements:

| Difference<br>Vertical | Gro | up I | Gro | · P value | |
|------------------------|-------|----------|-------|-----------|---------|
| Skeletal Measurements | MD | SD MD SD | | SD | r value |
| PP-SN angle | 0.31 | 0.91 | 0.17 | 0.27 | 0.66 |
| ANS-Me distance | 0.04 | 1.43 | -0.52 | 1.66 | 0.24 |
| MP-SN angle | -0.15 | 0.61 | -0.44 | 1.40 | 0.61 |

SD: standard deviation MD: mean difference



**Figure (62):** Bar chart showing comparison between both groups regarding vertical skeletal measurements.

#### B. Dental

# 1. Angular

#### a. Anteroposterior

#### • Group I:

In group I pretreatment records, post treatment records and difference between them regarding anteroposterior- angular- dental measurements were presented in table (21) and figure (63).

Comparison between pretreatment & post treatment records was performed by using Paired t-test which revealed insignificant difference between them in all measurements as P > 0.05 except U1-FHP and U5-FHP (Post was significantly higher than prerecord) as P < 0.05, as presented in table (21).

Table (21): Mean & standard deviation of pretreatment, post treatment records and difference between them regarding anteroposterior angular dental measurements in group I:

| Group I<br>Anteroposterior | Pı | Pre | | st | Difference | | |
|---|---|---|---|---|---|---|---|
| Angular Dental Measurements | M | SD | M | SD | MD | SD | P value |
| U1-NA | 25.83 | 9.57 | 26.27 | 10.17 | 0.44 | 1.88 | 0.437 |
| U1-FHP | 123.54 | 12.59 | 124.50 | 12.88 | 0.97 | 1.46 | 0.042* |
| U4-FHP | 102.14 | 9.64 | 103.24 | 11.70 | 1.10 | 4.80 | 0.444 |
| U5-FHP | 96.83 | 11.01 | 101.88 | 13.25 | 5.06 | 6.02 | 0.014* |
| U6-FHP | 94.43 | 8.90 | 89.70 | 9.02 | -4.72 | 9.69 | 0.119 |
| U7-FHP | 87.70 | 10.16 | 82.83 | 8.09 | -4.87 | 8.16 | 0.063 |

M: mean SD: standard deviation MD: mean difference



Figure (63): Bar chart showing mean of pretreatment, post treatment records and difference between them regarding anteroposterior angular dental measurements in group I.

#### • Group II:

In group II pretreatment records, post treatment records and difference between them regarding anteroposterior- angular- dental measurements were presented in table (22) and figure (64).

Comparison between pretreatment & post treatment records was performed by using Paired t-test which revealed insignificant difference between them in all measurements as P > 0.05 except U4-FHP and U5-FHP (Post records were significantly higher than prerecords), and U6-FHP (Post record was significantly lower than prerecord) as P < 0.05, as presented in table (22).

Table (22): Mean & standard deviation of pretreatment, post treatment records and difference between them regarding anteroposterior angular dental measurements in group II:

| Group II<br>Anteroposterior<br>Angular<br>Dental | pre | | po | post | | rence | P value |
|---|---|---|---|---|---|---|---|
| Measurements | M | SD | M | SD | MD | SD | |
| U1-NA | 16.88 | 4.94 | 17.05 | 5.79 | 0.18 | 0.85 | 0.67 |
| U1-FHP | 114.61 | 4.00 | 115.05 | 4.83 | 0.43 | 0.83 | 0.44 |
| U4-FHP | 105.26 | 5.30 | 109.68 | 4.81 | 4.42 | 5.18 | 0.034* |
| U5-FHP | 102.27 | 4.80 | 108.52 | 5.79 | 6.25 | 5.34 | 0.008* |
| U6-FHP | 97.77 | 1.80 | 84.23 | 9.21 | -13.54 | 8.61 | 0.002* |
| U7-FHP | 88.47 | 8.81 | 80.17 | 9.62 | -8.30 | 0.81 | 0.077 |

M: mean

SD: standard deviation

MD: mean difference



Figure (64): Bar chart showing pretreatment, post treatment records and difference between them regarding anteroposterior angular dental measurements in group II.

#### • Comparison between both groups:

Comparison between group I & II regarding difference between pretreatment & posttreatment records of anteroposterior angular dental measurements was performed by using Mann Whitney test which revealed insignificant difference between them regarding all measurements except U6-FHP (Group I was significantly higher than group II) as P < 0.05, as presented in table (23) and figure (65).

Table (23): Comparison between both groups regarding anteroposterior angular dental measurements:

| Difference<br>Anteroposterior | Gro | up I | Gro | Durke | |
|-------------------------------|-------|------|--------|-------|---------|
| Angular Dental Measurements | MD | SD | MD | SD | P value |
| U1-NA | 0.44 | 1.88 | 0.18 | 0.85 | 0.70 |
| U1-FHP | 0.97 | 1.46 | 0.43 | 0.83 | 0.33 |
| U4-FHP | 1.10 | 4.80 | 4.42 | 5.18 | 0.82 |
| U5-FHP | 5.06 | 6.02 | 6.25 | 5.34 | 0.61 |
| U6-FHP | -4.72 | 9.69 | -13.54 | 8.61 | 0.03* |
| U7-FHP | -4.87 | 8.16 | -8.30 | 0.81 | 0.16 |

SD: standard deviation MD: mean difference



Figure (65): Bar chart showing comparison between both groups regarding anteroposterior angular dental measurements.

#### b. Rotation

#### • Group I:

In group I pretreatment records, post treatment records and difference between them regarding rotation- angular- dental measurements were presented in table (24) and figure (66).

Comparison between pretreatment & post treatment records was performed by using Paired t-test which revealed insignificant difference between them in all measurements as P > 0.05 except U5-MSP and U7-MSP as there was a statistical significant difference as P < 0.05 (Post was significantly higher than prerecord), while in U6-MSP there was a highly statistical significant difference as P < 0.001 (Post was significantly higher than prerecord) as presented in table (24).

Table (24): Mean & standard deviation of pretreatment, post treatment records and difference between them regarding rotation angular dental measurements in group I:

| Group I<br>Rotation | Pre | | Post | | Diffe | | |
|---|---|---|---|---|---|---|---|
| Angular<br>Dental<br>Measurements | M | SD | M | SD | MD | SD | P value |
| U4-MSP | 71.89 | 6.73 | 74.95 | 6.62 | 3.06 | 8.70 | 0.248 |
| U5-MSP | 68.84 | 7.63 | 63.36 | 7.23 | -5.48 | 4.79 | 0.002* |
| U6-MSP | 32.38 | 6.45 | 50.50 | 10.29 | 18.12 | 8.35 | 0.000** |
| U7-MSP | 42.42 | 9.67 | 53.25 | 11.15 | 10.84 | 8.06 | 0.001* |

MD: mean difference

M: mean SD: standard deviation



**Figure (66):** Bar chart showing pretreatment, post treatment records and difference between them regarding rotation angular dental measurements in group I.

#### • Group II:

In group II pretreatment records, post treatment records and difference between them regarding rotation- angular- dental measurements were presented in table (25) and figure (67).

Comparison between pretreatment & post treatment records was performed by using Paired t-test which revealed insignificant difference between them in all measurements as P > 0.05 except U5-MSP and U6-MSP as there was a statistical significant difference as P < 0.05 (Post was significantly higher than prerecord), as presented in table (25).

Table (25): Mean & standard deviation of pretreatment, post treatment records and difference between them regarding rotation angular dental measurements in group II:

| Group II Rotation | pre | | post | | Difference | | P value |
|---|---|---|---|---|---|---|---|
| Angular<br>Dental<br>Meas urements | M | SD | M | SD | MD | SD | P value |
| U4-MSP | 74.75 | 5.74 | 75.51 | 7.01 | 0.76 | 7.22 | 0.761 |
| U5-MSP | 76.26 | 10.52 | 56.45 | 9.88 | -19.81 | 11.69 | 0.001* |
| U6-MSP | 32.33 | 6.82 | 51.46 | 19.53 | 19.13 | 19.26 | 0.018* |
| U7-MSP | 37.63 | 6.55 | 64.09 | 13.42 | 26.47 | 6.87 | 0.057 |

M: mean SD: standard deviation MD: mean difference



**Figure (67):** Bar chart showing mean of pretreatment, post treatment records and difference between them regarding rotation angular dental measurements in group II.

#### • Comparison between both groups:

Comparison between group I & II regarding difference between pretreatment & posttreatment records of rotation - angular dental measurements was performed by using Mann Whitney test which revealed insignificant difference between them regarding all measurements except U5-MSP (Group I was significantly higher than group II) as P < 0.05, as presented in table (26) and figure (68).

Table (26): Comparison between both groups regarding rotation angular dental measurements:

| Difference<br>Rotation | Gro | up I | Gro | D l | |
|-----------------------------|-------|------|--------|-------|---------|
| Angular Dental Measurements | MD | SD | MD | SD | P value |
| U4-MSP | 3.06 | 8.70 | 0.76 | 7.22 | 0.75 |
| U5-MSP | -5.48 | 4.79 | -19.81 | 11.69 | 0.009* |
| U6-MSP | 18.12 | 8.35 | 19.13 | 19.26 | 0.45 |
| U7-MSP | 10.84 | 8.06 | 26.47 | 6.87 | 0.06 |

SD: standard deviation

MD: mean difference



**Figure (68):** Bar chart showing comparison between both groups regarding rotation angular dental measurements.

#### c. Crown inclination

# • Group I:

In group I pretreatment records, post treatment records and difference between them regarding crown inclination- angular- dental measurements were presented in table (27) and figure (69).

Comparison between pretreatment & post treatment records was performed by using Paired t-test which revealed insignificant difference between them in all measurements as P > 0.05 except U4 and U5 as there was a statistically significant difference as P < 0.05 (Post was significantly higher than prerecord), as presented in table (27).

<u>Table (27): Mean & standard deviation of pretreatment, post treatment</u> <u>records and difference between them regarding crown inclination</u> angular dental measurements in group I:

| Group I<br>Crown | Pre | | Post | | Difference | | |
|---|---|---|---|---|---|---|---|
| Inclination Angular Dental Measurements | M | SD | M | SD | MD | SD | P value |
| U4 | 4.80 | 2.34 | 11.94 | 7.12 | 7.14 | 7.61 | 0.008* |
| U5 | 6.47 | 4.23 | 13.79 | 7.28 | 7.32 | 6.86 | 0.004* |
| U6 | 4.84 | 4.06 | 4.81 | 2.95 | -0.03 | 3.87 | 0.980 |
| U7 | 5.76 | 3.65 | 7.94 | 7.83 | 2.19 | 5.81 | 0.219 |

M: mean SD: standard deviation MD: mean difference



**Figure (69):** Bar chart showing mean of pretreatment, post treatment records and difference between them regarding crown inclination - angular dental measurements in group I.

#### • Group II:

In group II pretreatment records, post treatment records and difference between them regarding crown inclination- angular- dental measurements were presented in table (28) and figure (70).

Comparison between pretreatment & post treatment records was performed by using Paired t-test which revealed significant difference between them in all measurements as P < 0.05 except U5 as there was a statistical insignificant difference as P > 0.05 (Post was significantly higher than prerecord), as presented in table (28).

Table (28): Mean & standard deviation of pretreatment, post treatment records and difference between them regarding crown inclination - angular dental measurements in group II:

| Group II<br>Crown Inclination | pre | | post | | Difference | | P value |
|---|---|---|---|---|---|---|---|
| Angular<br>Dental Measurements | M | SD | M | SD | MD | SD | P value |
| U4 | 5.11 | 3.82 | 12.77 | 6.01 | 7.66 | 7.31 | 0.014* |
| U5 | 8.28 | 5.27 | 14.25 | 7.50 | 5.98 | 8.45 | 0.067 |
| U6 | 2.99 | 1.67 | 7.12 | 4.47 | 4.13 | 3.66 | 0.010* |
| U7 | 5.23 | 4.77 | 9.23 | 6.85 | 3.99 | 5.11 | 0.047* |

M: mean

SD: standard deviation

MD: mean difference



**Figure (70):** Bar chart showing mean of pretreatment, post treatment records and difference between them regarding crown inclination - angular dental measurements in group II.

# • Comparison between both groups:

Comparison between group I & II regarding difference between pretreatment & posttreatment records of crown inclination - angular dental measurements was performed by using Mann Whitney test which revealed insignificant difference between them regarding all measurements except U6 (Group I was significantly lower than group II) as P < 0.05, as presented in table (29) and figure (71).

<u>Table (29): Comparison between both groups regarding crown inclination</u> - angular dental measurements:

| Difference<br>Crown Inclination | Gro | up I | Gro | up II | P value |
|---------------------------------|-------|------|------|-------|---------|
| Angular Dental Measurements | MD | SD | MD | SD | r value |
| U4 | 7.14 | 7.61 | 7.66 | 7.31 | 0.86 |
| U5 | 7.32 | 6.86 | 5.98 | 8.45 | 0.71 |
| U6 | -0.03 | 3.87 | 4.13 | 3.66 | 0.04* |
| U7 | 2.19 | 5.81 | 3.99 | 5.11 | 0.27 |

SD: standard deviation MD: mean difference



**Figure (71):** Bar chart showing comparison between both groups regarding crown inclination - angular dental measurement.

#### 2. Linear

#### a. Anteroposterior

#### • Group I:

In group I pretreatment records, post treatment records and difference between them regarding anteroposterior- linear- dental measurements were presented in table (30) and figure (72). Comparison between pretreatment & post treatment records was performed by using Paired t-test which revealed insignificant difference between them in all measurements as P > 0.05 except U4-apex/S Ver and U5-apex/S Ver (Post was significantly higher than prerecord), MBc6/S Ver (Post was significantly lower than prerecord), as there was a statistical significant difference as P < 0.05, while in U5-tip/S Ver (Post was higher than pre),U6-apex/S Ver, MBc7/S Ver and U7-apex/S Ver (post was lower than pre) there was a highly statistical significant difference as P < 0.0001, as presented in table (30).
Table (30): Mean & standard deviation of pretreatment, post treatment records and difference between them regarding anteroposterior - linear dental measurements in group I:

| Group I<br>Anteroposterior | Pi | re | Po | st | Diffe | rence | |
|---|---|---|---|---|---|---|---|
| Linear<br>Dental<br>Measurements | M | SD | M | SD | MD | SD | P value |
| U1-tip/S Ver | 78.77 | 6.89 | 78.79 | 7.17 | 0.02 | 0.47 | 78.77 |
| U1-apex/SVer | 66.06 | 3.55 | 66.04 | 3.69 | -0.02 | 1.21 | 0.861 |
| L1-tip/S Ver | 72.47 | 3.99 | 71.31 | 4.58 | -1.16 | 2.50 | 0.948 |
| U4-tip/S Ver | 61.06 | 3.77 | 62.11 | 3.94 | 1.06 | 1.17 | 0.124 |
| U4-apex/S Ver | 57.08 | 3.56 | 59.67 | 3.11 | 2.59 | 1.64 | 0.010* |
| U5-tip/S Ver | 54.68 | 3.61 | 56.08 | 3.71 | 1.40 | 1.00 | 0.000** |
| U5-apex/S Ver | 52.57 | 2.51 | 54.42 | 2.71 | 1.86 | 1.55 | 0.001* |
| MBc6/S Ver | 48.60 | 3.53 | 44.82 | 3.35 | -3.78 | 1.31 | 0.002* |
| U6-apex/S Ver | 47.70 | 3.06 | 44.92 | 2.83 | -2.78 | 1.64 | 0.000** |
| MBc7/S Ver | 37.47 | 3.57 | 34.21 | 3.32 | -3.26 | 1.55 | 0.000** |
| U7-apex/S Ver | 37.79 | 2.65 | 35.29 | 3.44 | -2.50 | 2.45 | 0.000** |
| overjet | 6.30 | 3.52 | 7.48 | 5.46 | 1.19 | 2.43 | 0.311 |



In group II pretreatment records, post treatment records and difference between them regarding anteroposterior- linear- dental measurements were presented in table (31) and figure (73).

Comparison between pretreatment & post treatment records was performed by using Paired t-test which revealed insignificant difference between them in all measurements as P >0.05 except U4-apex/S Ver U5-tip/S Ver, U5-apex/S Ver (Post was significantly higher than prerecord and MBc6/S Ver , U6-apex/S Ver , MBc7/S Ver & U7-apex/S Ver (Post was significantly lower than prerecord), as there was a statistical significant difference as P < 0.05, , as presented in table (31).

Table (31): Mean & standard deviation of pretreatment, post treatment records and difference between them regarding anteroposterior - linear dental measurements in group II:

| Group II<br>Anteroposterior | pı | re | po | ost | Diffe | rence | n I. |
|---|---|---|---|---|---|---|---|
| Linear<br>Dental<br>Meas urements | M | SD | M | SD | MD | SD | P value |
| U1-tip/S Ver | 76.89 | 2.86 | 77.48 | 2.99 | 0.59 | 0.13 | 0.12 |
| U1-apex/ S Ver | 67.13 | 3.09 | 67.56 | 3.18 | 0.43 | 0.08 | 0.25 |
| L1-tip/S Ver | 72.48 | 3.32 | 71.93 | 4.20 | -0.54 | 1.61 | 0.342 |
| U4-tip/S Ver | 63.21 | 3.81 | 64.32 | 4.43 | 1.11 | 1.76 | 0.095 |
| U4-apex/S Ver | 57.90 | 3.53 | 59.69 | 2.68 | 1.79 | 1.19 | 0.002* |
| U5-tip/S Ver | 56.43 | 3.58 | 58.31 | 3.87 | 1.88 | 1.49 | 0.005* |
| U5-apex/S Ver | 53.48 | 2.83 | 54.85 | 2.27 | 1.37 | 1.58 | 0.031* |
| MBc6/S Ver | 50.55 | 3.53 | 46.04 | 5.61 | -4.51 | 3.39 | 0.004* |
| U6-apex/S Ver | 48.06 | 3.97 | 45.94 | 5.17 | -2.12 | 2.52 | 0.035* |
| MBc7/S Ver | 39.93 | 3.98 | 34.61 | 5.39 | -5.32 | 3.62 | 0.002* |
| U7-apex/S Ver | 39.18 | 3.01 | 36.79 | 2.75 | -2.40 | 0.98 | 0.000** |
| overjet | 4.46 | 1.63 | 5.31 | 1.99 | 0.85 | 1.25 | 0.074 |



Figure (73): Bar chart showing mean of pretreatment, post treatment records and difference between them regarding anteroposterior linear dental measurements in group II.

Comparison between group I & II regarding difference between pretreatment & posttreatment records of anteroposterior - linear dental measurements was performed by using Mann Whitney test which revealed insignificant difference between them regarding all measurements except U1-tip/S Ver (Group I was significantly lower than group II) as P < 0.05, as presented in table (32) and figure (74).

<u>Table (32): Comparison between both groups regarding anteroposterior - linear dental measurements:</u>

| Difference<br>Anteroposterior | Gro | up I | Gro | up II | · P value |
|-------------------------------|-------|------|-------|-------|-----------|
| Linear<br>Dental Measurements | MD | SD | MD | SD | P value |
| U1-tip/S Ver | 0.02 | 0.47 | 0.59 | 0.13 | 0.002* |
| U1-apex/ S Ver | -0.02 | 1.21 | 0.43 | 0.08 | 0.28 |
| L1-tip/S Ver | -1.16 | 2.50 | -0.54 | 1.61 | 1 |
| U4-tip/S Ver | 1.06 | 1.17 | 1.11 | 1.76 | 0.97 |
| U4-apex/S Ver | 2.59 | 1.64 | 1.79 | 1.19 | 0.31 |
| U5-tip/S Ver | 1.40 | 1.00 | 1.88 | 1.49 | 0.71 |
| U5-apex/S Ver | 1.86 | 1.55 | 1.37 | 1.58 | 0.71 |
| MBc6/S Ver | -3.78 | 1.31 | -4.51 | 3.39 | 0.8 |
| U6-apex/S Ver | -2.78 | 1.64 | -2.12 | 2.52 | 1 |
| MBc7/S Ver | -3.26 | 1.55 | -5.32 | 3.62 | 0.12 |
| U7-apex/S Ver | -2.50 | 2.45 | -2.40 | 0.98 | 0.86 |
| overjet | 1.19 | 2.43 | 0.85 | 1.25 | 0.75 |



linear dental measurements.

#### b. Vertical

### • Group I:

In group I pretreatment records, post treatment records and difference between them regarding vertical- linear- dental measurements were presented in table (33) and figure (75).

Comparison between pretreatment & post treatment records was performed by using Paired t-test which revealed significant difference between them in all measurements as P < 0.05 except overbite as there was insignificant difference between pre & post as P > 0.05. In U1-tip/PP, pre was significantly lower than post, while in U4-tip/PP, U5-tip/PP, MBc6/PP, MBc7/PP and L1-tip/PP pre was significantly higher than post as P < 0.05, as presented in table (33).

Table (33): Mean & standard deviation of pretreatment, post treatment records and difference between them regarding vertical - linear dental measurements in group I:

| Group I<br>Vertical | Pı | Pre | | st | Diffe | rence | |
|---|---|---|---|---|---|---|---|
| Linear<br>Dental<br>Measure ments | M | SD | M | SD | MD | SD | P value |
| U1-tip/PP | 27.68 | 3.67 | 27.86 | 3.67 | 0.18 | 0.52 | 0.005* |
| U4-tip/PP | 25.79 | 3.18 | 25.10 | 3.00 | -0.69 | 0.56 | 0.001* |
| U5-tip/PP | 25.25 | 2.82 | 24.56 | 3.01 | -0.70 | 0.63 | 0.001* |
| MBc6/PP | 23.90 | 2.50 | 22.75 | 2.75 | -1.15 | 0.88 | 0.003* |
| MBc7/PP | 21.43 | 2.81 | 20.77 | 3.24 | -0.65 | 0.91 | 0.001* |
| L1-tip/PP | 24.45 | 3.73 | 23.63 | 5.55 | -0.82 | 2.67 | 0.008* |
| overbite | 3.23 | 1.14 | 4.23 | 2.57 | 1.00 | 2.68 | 0.119 |



Figure (75): Bar chart showing mean of pretreatment, post treatment records and difference between them regarding vertical linear dental measurements in group I.

In group II pretreatment records, post treatment records and difference between them regarding vertical- linear- dental measurements were presented in table (34) and figure (76).

Comparison between pretreatment & post treatment records was performed by using Paired t-test which revealed insignificant difference between them in all measurements as P > 0.05 except U4-tip/PP, MBc6/PP & MBc7/PP as Pre was significantly higher than post as P < 0.05., as presented in table (34).

Table (34): Mean & standard deviation of pretreatment, post treatment records and difference between them regarding vertical - linear dental measurements in group II:

| Group II<br>Vertical | pre | | po | ost | Diffe | rence | |
|---|---|---|---|---|---|---|---|
| Linear<br>Dental<br>Measurements | M | SD | M | SD | M | SD | P value |
| U1-tip/PP | 27.78 | 3.27 | 28.05 | 3.19 | 0.27 | -0.09 | 0.16 |
| U4-tip/PP | 25.98 | 2.93 | 25.25 | 3.13 | -0.73 | 0.86 | 0.036* |
| U5-tip/PP | 25.21 | 3.05 | 24.76 | 3.62 | -0.45 | 1.36 | 0.352 |
| MBc6/PP | 24.00 | 3.28 | 22.47 | 3.13 | -1.53 | 1.21 | 0.005* |
| MBc7/PP | 22.00 | 3.65 | 20.11 | 3.72 | -1.88 | 1.83 | 0.015* |
| L1-tip/PP | 24.74 | 4.08 | 24.18 | 4.37 | -0.56 | 1.79 | 0.374 |
| overbite | 3.56 | 2.61 | 4.67 | 2.43 | 1.11 | 1.47 | 0.053 |

M: mean SD: standard deviation

MD: mean difference



difference between them regarding vertical linear dental measurements in group II. Figure (76): Bar chart showing mean of pretreatment, post treatment records and

Comparison between group I & II regarding difference between pretreatment & posttreatment records of vertical - linear dental measurements was performed by using Mann Whitney test which revealed insignificant difference between them regarding all measurements, as presented in table (35) and figure (77).

<u>Table (35): Comparison between both groups regarding vertical - linear dental measurements:</u>

| Difference<br>Vertical | Gro | up I | Grou | ıp II | P value |
|----------------------------|-------|------|-------|-------|---------|
| Linear Dental Measurements | MD | SD | MD | SD | P Value |
| U1-tip/PP | 0.18 | 0.52 | 0.27 | -0.09 | 0.61 |
| U4-tip/PP | -0.69 | 0.56 | -0.73 | 0.86 | 0.81 |
| U5-tip/PP | -0.70 | 0.63 | -0.45 | 1.36 | 0.86 |
| MBc6/PP | -1.15 | 0.88 | -1.53 | 1.21 | 0.81 |
| MBc7/PP | -0.65 | 0.91 | -1.88 | 1.83 | 0.11 |
| L1-tip/PP | -0.82 | 2.67 | -0.56 | 1.79 | 0.65 |
| overbite | 1.00 | 2.68 | 1.11 | 1.47 | 0.27 |

SD: standard deviation

MD: mean difference



Figure (77): Bar chart showing comparison between both groups regarding vertical linear dental measurements

#### c. Transverse

#### • Group I:

In group I pretreatment records, post treatment records and difference between them regarding transverse- linear- dental measurements were presented in table (36) and figure (78).

Comparison between pretreatment & post treatment records was performed by using Paired t-test which revealed significant difference between them in all measurements as P < 0.05 except U4 as there was insignificant difference between pre & post as P > 0.05. In U5, there was a statistically significant difference as P < 0.05 (pre was significantly lower than post), while in U6 and U7 there was a highly statistical significant difference as P < 0.001 (pre was significantly lower than post), as presented in table (36).

Table (36): Mean & standard deviation of pretreatment, post treatment records and difference between them regarding transverse - linear dental measurements in group I:

| Group I<br>Transverse | Pre | | Po | Post | | rence | P value |
|---|---|---|---|---|---|---|---|
| Linear<br>Dental Measurements | M | SD | M | SD | MD | SD | r value |
| U4 | 16.80 | 2.01 | 18.55 | 2.03 | 1.75 | 1.36 | 0.438 |
| U5 | 18.83 | 2.06 | 20.84 | 1.94 | 2.01 | 1.11 | 0.001* |
| U6 | 21.96 | 2.21 | 23.39 | 2.06 | 1.43 | 0.98 | 0.000** |
| U7 | 24.50 | 2.55 | 25.45 | 2.50 | 0.95 | 1.01 | 0.000** |

M· mean

SD: standard deviation

MD: mean difference



**Figure (78):** Bar chart showing mean of pretreatment, post treatment records and difference between them regarding transverse - linear dental measurements in group I.

In group II pretreatment records, post treatment records and difference between them regarding transverse- linear- dental measurements were presented in table (37) and figure (79).

Comparison between pretreatment & post treatment records was performed by using Paired t-test which revealed insignificant difference between them in all measurements as P < 0.05, as presented in table (37).

Table (37): Mean & standard deviation of pretreatment, post treatment records and difference between them regarding transverse - linear dental measurements in group II:

| Group II<br>Transverse | pre | | po | post | | rence | P value |
|---|---|---|---|---|---|---|---|
| Linear<br>Dental Measurements | M | SD | M | SD | M | SD | r value |
| U4 | 17.45 | 2.12 | 18.04 | 2.02 | 0.60 | 1.95 | 0.387 |
| U5 | 20.04 | 1.82 | 20.80 | 2.00 | 0.76 | 1.59 | 0.188 |
| U6 | 23.01 | 1.76 | 23.66 | 1.35 | 0.65 | 1.15 | 0.130 |
| U7 | 25.04 | 2.14 | 25.06 | 1.80 | 0.02 | 2.30 | 0.984 |



**Figure (79):** Bar chart showing mean of pretreatment, post treatment records and difference between them regarding transverse - linear dental measurements in group II.

Comparison between group I & II regarding difference between pretreatment & posttreatment records of transverse — linear dental measurements was performed by using Mann Whitney test which revealed insignificant difference between them regarding all measurements except U5 (Group I was significantly higher than group II) as P < 0.05, as presented in table (38) and figure (80).

<u>Table (38): Comparison between both groups regarding transverse - linear dental measurements:</u>

| Difference<br>Transverse | Gro | up I | Gro | D lu | |
|-------------------------------|------|------|------|------|---------|
| Linear<br>Dental Measurements | MD | SD | MD | SD | P value |
| U4 | 1.75 | 1.36 | 0.60 | 1.95 | 0.19 |
| U5 | 2.01 | 1.11 | 0.76 | 1.59 | 0.04* |
| U6 | 1.43 | 0.98 | 0.65 | 1.15 | 0.09 |
| U7 | 0.95 | 1.01 | 0.02 | 2.30 | 0.31 |

SD: standard deviation

MD: mean difference



Figure (80): Bar chart showing comparison between both groups regarding transverse -linear dental measurements.

#### C. Soft tissue

## • Group I:

In group I pretreatment records, post treatment records and difference between them regarding soft tissue measurements were presented in table (39) and figure (81,82).

Comparison between pretreatment & post treatment records was performed by using Paired t-test which revealed insignificant difference between them in all measurements as P > 0.05, as presented in table (39).

Table (39): Mean & standard deviation of pretreatment, post treatment records and difference between them regarding soft tissue measurements in group I:

| Group I<br>Soft tissue | P | Pre | | Post | | rence | Dwalna |
|---|---|---|---|---|---|---|---|
| Me asure ments | M | SD | M | SD | MD | SD | P value |
| Ls/E-line distance | 2.72 | 1.27 | 2.81 | 0.74 | 0.10 | 0.70 | 0.643 |
| Li/E-line distance | 2.40 | 1.58 | 2.05 | 1.46 | -0.36 | 0.96 | 0.226 |
| NLA angle | 97.44 | 12.44 | 98.61 | 13.17 | 1.17 | 3.37 | 0.253 |



**Figure (81):** Bar chart showing mean of pretreatment, post treatment records and difference between them regarding Ls/E-line distance & Li/E-line distance in group I.



Figure (82): Bar chart showing Mean of pretreatment, post treatment records and difference between them regarding NLA angle in Group I.

In group II pretreatment records, post treatment records and difference between them regarding soft tissue measurements were presented in table (40) and figure (83,84).

Comparison between pretreatment & post treatment records was performed by using Paired t-test which revealed insignificant difference between them in all measurements as P > 0.05, as presented in table (40).

Table (40): Mean & standard deviation of pretreatment, post treatment records and difference between them regarding soft tissue measurements in group II:

| Group II | Pi | Pre | | Post | | rence | P value |
|---|---|---|---|---|---|---|---|
| Soft tissue<br>Measurements | M | SD | M | SD | MD | SD | P value |
| Ls/E-line distance | 3.61 | 2.78 | 3.22 | 2.14 | -0.40 | 2.34 | 0.625 |
| Li/E-line distance | 2.86 | 2.00 | 2.23 | 1.74 | -0.63 | 2.13 | 0.403 |
| NLA angle | 105.30 | 9.52 | 105.91 | 6.47 | 0.61 | 3.98 | 0.656 |



**Figure (83):** Bar chart showing mean of pretreatment, post treatment records and difference between them regarding Ls/E-line distance & Li/E-line distance in group II.



**Figure (84):** Bar chart showing mean of pretreatment, post treatment records and difference between them regarding Mean of NLA angle in Group II.

Comparison between group I & II regarding difference between pretreatment & posttreatment records of soft tissue measurements was performed by using Mann Whitney test which revealed insignificant difference between them regarding all measurements, as presented in table (41) and figure (85).

<u>Table (41): Comparison between both groups regarding soft tissue</u> measurements:

| Difference | Gro | up l | Gro | P value | |
|--------------------------|-------|------|-------|---------|---------|
| Soft tissue Measurements | MD | SD | MD | SD | P value |
| Ls/E-line distance | 0.10 | 0.70 | -0.40 | 2.34 | 0.75 |
| Li/E-line distance | -0.36 | 0.96 | -0.63 | 2.13 | 0.71 |
| NLA angle | 1.17 | 3.37 | 0.61 | 3.98 | 0.35 |



**Figure (85):** Bar chart showing comparison between both groups regarding soft tissue measurement